CLINICAL TRIAL: NCT06731868
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Safety, Tolerability, Preliminary Efficacy and Pharmacokinetic Characteristics of Multiple Doses of LPM3770164 Sustained-release Tablets in Patients With Tardive Dyskinesia
Brief Title: Safety and Efficacy of LPM3770164 Sustained-release Tablets in Patients With Tardive Dyskinesia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY03015/CT-CHN-204
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Tardive Dyskinesia (TD)
MeSH Terms: conditions — Tardive Dyskinesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LPM3770164 sustained release tablet 5 mg (Experimental)
  Interventions: Drug: LPM3770164 sustained release tablet 5 mg
- LPM3770164 sustained release tablet 10 mg (Experimental)
  Interventions: Drug: LPM3770164 sustained release tablet 10 mg
- LPM3770164 sustained release tablet 20 mg (Experimental)
  Interventions: Drug: LPM3770164 sustained release tablet 20 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: LPM3770164 sustained release tablet simulant

INTERVENTIONS:
Drug: LPM3770164 sustained release tablet 5 mg — LPM3770164 sustained release tablet once daily oral dosage at 5 mg for 6 weeks
  Other Names: LY03015
  Arms: LPM3770164 sustained release tablet 5 mg
Drug: LPM3770164 sustained release tablet 10 mg — LPM3770164 sustained release tablet once daily oral dosage at 10 mg for 6 weeks.
  Other Names: LY03015
  Arms: LPM3770164 sustained release tablet 10 mg
Drug: LPM3770164 sustained release tablet 20 mg — LPM3770164 sustained release tablet once daily oral dosage at 20 mg for 6 weeks.
  Other Names: LY03015
  Arms: LPM3770164 sustained release tablet 20 mg
Drug: LPM3770164 sustained release tablet simulant — LPM3770164 sustained release tablet simulant once daily oral for 6 weeks.
  Other Names: placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled parallel-group trial to evaluate the safety, tolerability, preliminary efficacy and PK characteristics of multiple doses of LPM3770164 sustained-release tablets in TD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who voluntarily participate in and sign the informed consent form;
2. Male or female subjects aged ≥ 18 years and < 65 years;
3. Body mass index (BMI) 18.5 ~ 38.0 kg/m2 (including boundary value);
4. Subjects with a past diagnosis of schizophrenia, schizoaffective disorder, bipolar and related disorders, depressive disorders based on medical history, and stable for at least 1 month;
5. Subjects who have been diagnosed with medication-induced TD, and whose symptoms have lasted for at least 3 months according to the DSM-5; and TD is assessed as moderate or severe (AIMS Item 8 score ≥3);
6. Medications for schizophrenia, schizoaffective disorder, bipolar and related disorders, depressive disorders and extrapyramidal reactions should be kept dose stable for at least 1 month (benzodiazepines should stable at least 14 days, Long-acting injection should stable for at least 3 months);
7. Females of childbearing potential have a negative pregnancy test. Male and female patients of childbearing potential and their spouses/partners agree to not plan to become pregnant (including the plan for sperm and egg donation) and to use effective contraceptive measures throughout the study and for at least 1 month after the last dose of the study drug.

Exclusion Criteria:

1. Has comorbid abnormal involuntary movement(s) that is more prominent than TD as judged by the investigator;
2. Has Simpson-Angus Scale (SAS) score≥ 3 on two or more items other than items 8 and 10;
3. Currently in the acute phase of mental disorder or severe psychiatric symptoms, unable to cooperate with the treatment and assessment, as judged by the investigator;
4. Has a history of suicide attempt or Question 4 or Question 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) as "Yes" within the past 6 months;
5. Has a history of neuroleptic-related malignant syndrome;
6. Has diagnosed with malignant tumor within 3 years before randomization;
7. Has a history of long QT syndrome or tachyarrhythmia within 3 years before randomization;
8. Electrocardiogram QTcF > 450 ms, or other clinically significant ECG findings in the opinion of the investigator;
9. Patients with significant abnormal liver and kidney function indicators, meeting any of the following criteria: serum creatinine > 1.5 × upper limit of normal (ULN); serum alanine transaminase (ALT) or aspartate transaminase (AST) > 2.5 × ULN; total bilirubin > 1.5 × ULN;
10. Has active, severe and unstable cerebrovascular, liver, kidney, endocrine, cardiovascular, gastrointestinal, respiratory, or metabolic disorders within 30 days prior to screening, in the judgment of the investigator, would interfere with the patient's ability to participate in the trial;
11. Any surgical condition or condition that may significantly affect the absorption, distribution, metabolism and excretion of the drug, or may pose a hazard to the subjects participating in the trial, such as but not limited to history of gastrointestinal surgery (gastrectomy, gastrointestinal anastomosis, intestinal resection, etc.), urinary tract obstruction or dysuria, gastroenteritis, gastrointestinal ulcers, gastrointestinal bleeding;
12. Has a known history of allergy to any component of the investigational product or similar drugs, or allergic constitution;
13. Has a positive human immunodeficiency virus antibody (HIV-Ab) and syphilis;
14. Has a positive urine drug screen;
15. Patients diagnosed with substance-related and addictive disorders (except tobacco- or caffeine-related disorders) within 6 months prior to the screening visit;
16. Has participated in any clinical trials of drugs (excluding vitamins and minerals) within 3 months prior to the screening visit;
17. Patients who previously received deep brain stimulation (DBS), or received electroconvulsive therapy (ECT) or other physical therapy within 1 month prior to the screening visit;
18. Patients who use of strong inducers or inhibitors of CYP3A4 within 14 days or 5 half-lives, whichever is longer, prior to randomization;
19. Known history of a nonresponder to tetrabenazine, deutetrabenazinen, or valbenazine for the treatment of TD;
20. Patients who have been injected with botulinum toxin in the past 3 months;
21. Patients who have used the prohibited drugs in the past 1 month;
22. Nursing mothers;
23. For patients with schizophrenia and schizoaffective disorder, has a total PANSS score > 80, and/or a total CDSS score > 10;
24. For patients with bipolar and related disorders or depressive disorders, has a history of rapid cycling, or a total MADRS score > 22, or a total YMRS score > 12;
25. Other conditions judged by the investigator as unsuitable for participating in the trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse event | From baseline to Week 8
  Number of participants with treatment-emergent adverse event will be summarized by Group, System Organ Classification (SOC), Preferred Term (PT), severity and the relationship with treatment.
Change in Abnormal Involuntary Movement Scale (AIMS) Dyskinesia Total Score | From baseline to Week 8
  Severity of TD symptoms assessed by AIMS dyskinesia total score (sum of items 1 through 7), as assessed by blinded AIMS raters. The AIMS Total Dyskinesia Score rates a total of 7 items, rating involuntary movement from 0 (no dyskinesia) to 4 (severe dyskinesia). Items 1 through 7 include facial and oral movements (Items 1-4), extremity movements (Items 5-6), and trunk movements (Item 7). The AIMS dyskinesia total score for Items 1-7 ranges from 0 to 28; a higher score reflects increased severity.

SECONDARY OUTCOMES:
The proportion of subjects who have a 50% improvement in AIMS Dyskinesia Total Score | From baseline to Week 8
Clinical Global Impression - Global Improvement of TD (CGI-TD) | From Week 2 to Week 8
Patient Global Impression of Change (PGIC) | From Week 2 to Week 8
Maximum observed concentration (Cmax) | From predose to 24 hours of day 1
Area Under the Curve from time 0 to 24 hours of day 1 (AUC0-24h) | From predose to 24 hours of day 1
Concentration at the end of the dosing interval at steady state (Cτ,ss) | Predose on Day 14±2, Day 28±2 and Day 42±2

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China